CLINICAL TRIAL: NCT02382523
Title: Impact of Acthar on Proteinuria and Disease Progression in IgA Nephropathy Patients With Nephrotic Range Proteinuria
Brief Title: Acthar on Proteinuria in IgA Nephropathy Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: There were no subjects enrolled locally on this study since it opened. Local IRB closure has been requested.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Sheikh-Hamad, Professor (Medicine-Nephrology), Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32884 Acthar IgA Nephropathy
Record Dates: First submitted 2015-01-09; First posted 2015-03-06 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: IgA Nephropathy; Proteinuria
Keywords: acthar; proteinuria; IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acthar injection 2 times per week (Experimental): Acthar 80 unit injection 2 times a week
  Interventions: Drug: Acthar 80 unit injection
- Acthar injection 3 times per week (Experimental): Acthar 80 unit injection 3 times a week
  Interventions: Drug: Acthar 80 unit injection

INTERVENTIONS:
Drug: Acthar 80 unit injection — Subjects not responding after 3 months of therapy (increasing creatinine; proteinuria not lower by 30%), will continue therapy at a dose 120 U SC x2/wk. Treatment will be discontinued if improvement is not observed 6 months after initiation of therapy.
  If partial remission is achieved with Acthar 80 U SC x2/wk or x3/wk then Acthar will be increased to 120 U SCx2/wk; if remission is achieved, treatment will be continued at this dose for a total of 12 months; otherwise, if response is not observed after 3 months of treatment with the higher dose, we will resume therapy with the original dose/schedule. We will check anti-ACTH antibodies in non-responders.
  If relapse occurs during the follow-up period, a 6 month treatment with Acthar at 120 U SC x2/wk will be started (not for partial responders), and the response will be assessed.
  Other Names: H.P. Acthar gel

SUMMARY:
IgA nephropathy occurs when IgA-a protein that helps the body fight infections-settles in the kidneys. IgA deposits may cause the kidneys to leak blood and sometimes protein in the urine. Proteinuria (abnormal amounts of protein in urine) can be a sign of kidney damage. Current treatments for IgA nephropathy is limited to Angiotensin Converting Enzyme (ACE) inhibitor medications with fish oil. ACE Inhibitors, also called ACEI medications, slows the angiotensin converting enzyme so that blood vessels can be relaxed.

This study involves the study drugs, Acthar and Lisinopril (an ACEI medication routinely given for high blood pressure).

In previous clinical studies, some subjects with IgA nephropathy have experienced reductions in proteinuria with consistent use of Acthar. Acthar is approved by the Food and Drug Administration (FDA) and used to treat patients with proteinuria.

The purpose is to study the safety and effectiveness of the study drug Acthar given at different doses.

DETAILED DESCRIPTION:
Participation in this study may last up to 2 years (from first visit to final visit) and includes 10 study visits and 8 phone calls.

Subjects will be randomly assigned to one of two treatment groups:

Group A will receive Acthar 80 unit injection 2 times per week or

Group B will receive Acthar 80 unit injection 3 times per week

All participants will be prescribed Lisinopril (10mg per day or higher depending on your blood pressure) as part of regular care for their condition. If they are already on another ACEI, Lisinopril will be prescribed. If subjects are unable to tolerate Lisinopril or other ACEI medications, an angiotensin receptor blocker (ARB) will be prescribed. ARBs are another type of medication that also helps relax blood vessels if subjects cannot tolerate ACEI medications.

Regardless of which treatment group subjects are assigned,everyone will self-inject the study drug using a subcutaneous (SC) injection under the skin using a needle and syringe. Subjects will be trained on the proper technique to be used for each injection before taking study drug home. Enough of the study drug will be given to take home (based on which group the subject is in) to administer until they are seen in 3 months for their next study visit.

Blood samples will be taken for lab tests at each visit and biomarkers (Screening Visit and Visit 9). Women of childbearing potential will also have a pregnancy test done. Approximately 4 teaspoons of blood will be drawn for the Screening Visit and Visit 9.

Subjects must fast at least 8 hours prior to the blood draw.

The following study procedures will be performed:

SCREENING VISIT:

* Informed consent will be obtained;
* Inclusion/exclusion criteria will be assessed, demographics and medical history will be collected (including PCR and urinalysis results as these tests are routinely done as part of regular care);
* Pregnancy test if subject is a female of child bearing potential;
* Physical exam;
* Height/Weight collected;
* Vital signs will be obtained. Blood pressure will be recorded.
* Blood samples collected for study specific tests (aldosterone and cortisol) (approximately 2 teaspoons) and biomarkers (approximately 2 teaspoons). No more than approximately 4 teaspoons will be collected at this study visit;

Subjects who do not meet eligibility criteria during the initial screening attempt will be permitted to rescreen 2 times, for a total of 3 screening attempts. Rescreen subjects must first be registered as screen failed in the CTMS system and subsequently registered as a rescreen subject. Once the subject is registered as rescreened, all screening procedures will need to be repeated.;The exact time interval of each re-screen would be at the discretion of the investigator. Completion of rescreen would be no greater than 6 months from the initial screening date.

VISIT 1 (BASELINE, DAY 0)

* Pregnancy test if subject is a female of child bearing potential
* The first study drug dose in the clinic under the supervision of the study staff. Subject will remain at the clinic for at least 1 hour for monitoring of any allergic reaction.
* Subjects will receive enough study drug (8 for those dosing twice a week and 11 for those dosing three times a week) to take home until their next visit in 3 months. Subjects will also receive a dosing diary to keep track of each dose taken and any side effects they may feel. Subjects will bring dosing diary with them to each study visit on Visits 2-5.

A member of the study staff will also call subjects once a week for the first 4 weeks after starting study drug (Visit 1) to make sure they are taking the study drug as required, completing the dosing diary, if they are taking any other medications and if they are experiencing any side effects. There will be 4 phone calls between Visit 1 and Visit 2.

VISITS 2-5 ONLY (MONTHS 3, 6, 9, 12)

* Dosing diary is collected
* Study medication accountability is recorded.
* Pregnancy test if subject is a female of child bearing potential
* Acthar medication is dispensed (Visits 2-4 only)
* Kidney biopsy performed - Visit 5 only

Kidney biopsy procedure:

Subjects will have to go to nearby hospital within 1 week of completing Visit 5 to have this outpatient procedure done. Subjects will be asked to lie on their stomach face down with a pillow under their rib cage for at least 20 to 30 minutes. Ultrasound may be used to find the proper biopsy site. A local numbing medicine (anesthetic) will be injected under their skin near the biopsy area.

The hospital staff will make a tiny cut in the skin and insert a biopsy needle into the area and to the surface of the kidney. Subjects will be asked to take a deep breath and hold breath as a thin needle is passed through the skin into the kidney. Inside the needle is a sharp edge that will remove small pieces of the kidney. The biopsy needle will then be withdrawn, and pressure will be applied to the biopsy site to stop the minor bleeding that usually occurs after the biopsy. After the procedure, a bandage will be applied to the biopsy site.

The hospital staff will give subject numbing or pain medicines as needed.

VISITS 2-9 (MONTHS 3, 6, 9, 12, 15, 18, 24)

* Inclusion/exclusion criteria will be assessed, demographics and medical history will be collected;
* Physical exam;
* Height/Weight collected;
* Vital signs will be obtained. Blood pressure will be recorded.
* Blood samples collected for study specific tests (aldosterone and cortisol) (approximately 2 teaspoons). Biomarkers (approximately 2 teaspoons) will also be collected at Visit 9. No more than approximately 4 teaspoons will be collected at Visit 9;

After Visit 2, a member of the study staff will continue to call you about every 1 ½ months to make sure subjects are taking the study drug as required, if subjects are taking any other medications and if they are experiencing any side effects. There will be 4 more phone calls that will occur between Visit 2-3, Visit 3-4, Visit 4-5 and Visit 5-6. Subjects will receive a total of 8 phone calls during this study.

The total amount of blood collected over the course of this study is no more than approximately 38 teaspoons.

Treatment with the study drugs will continue for the first 12 months of participation in this study. If subjects do not respond after 3 months of treatment or only partially respond to the treatment, dosage may be increased (up to 120 unit injections twice a week for 3 months). If subjects still do not respond at the increased dose, the study drug will be discontinued after another 3 months of treatment.

If subjects respond to the treatment during the 12 months of treatment but then their response goes away during the follow up period, they will be placed back on study drug for an additional 6 months.

If, for any reason, the study drug is stopped before the last treatment visit, subjects will be asked to come into the clinic to complete study procedures. Subjects will be asked to have all end-of-study testing done for safety.

Acthar cannot be abruptly stopped and must be gradually lessened. Except if subjects are experiencing an allergic reaction, the drug will be administered at half the dose for 1 week, then ¼ dose for another week, then stopped.

If subjects are on insulin or other oral antidiabetic medications, Acthar may decrease glucose (sugar) tolerance. This may result in an increase blood sugar. Subjects will be asked to let the study doctor know if they are on these medications to discuss glucose monitoring and a plan on how to keep taking these medications while on Acthar and what to do if they experience an increase in blood sugar.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study specific procedures
2. Male and females aged 18 years and older
3. BMI 40 kg/m2 or less
4. History of nephrotic syndrome due to IgA (confirmed from renal biopsy performed within last 5 years)
5. Protein to creatinine (PCR) ratio 2.5 g/g or more (spot urine)
6. Estimated GFR (eGFR) greater than 30 mL/min/1.73/m2 (as calculated using the abbreviated Modification of Diet in Renal Disease [MDRD] equation as per http://www.kidney.org/professionals/kdoqi/gfr_calculator.cfm).
7. Any prior course of therapy with (but not within the last 3 months): steroids, cyclophosphamide, chlorambucil, cyclosporine or tacrolimus ). If, after f/u period, it was determined that subject did not achieve a complete or partial response, subject will be eligible for this study.
8. Antihypertensive treatment including use of Angiotensin-converting enzyme inhibitors (ACEI) and/or Angiotensin receptor blockers (ARB):

   * Unless there is a history of intolerance to ACEI or ARB therapy, the subject must be treated with at least one of these agents,
   * Treatment with ACEI and/or ARB for 3 months or more prior to Visit 1, with stable maintenance dose(s) for 30 days or more prior to Visit 1,
   * If treated with other antihypertensive therapies, treatment duration of 30 days or more and stable maintenance dose for 7 days or more prior to Visit 1; and
9. Blood pressure determined by the average of 3 or more seated readings taken 5 minutes or more apart at Visit 1:

   * Mean systolic blood pressure 140 mmHg or less and
   * Mean diastolic blood pressure 80 mmHg or less.
10. Subjects must have the following laboratory results for study inclusion:

    * Hemoglobin 9 g/dL or more
    * Platelets 100 X 10^3 cells/mu-L
    * AST 2x ULN or less
    * ALT 2x ULN or less
    * Total bilirubin 2x ULN or less
    * HgbA1c less than 6.5%

Exclusion Criteria:

1. Inability or refusal to give informed consent
2. Unwillingness to receive or intolerant of SC injections of study medication
3. Use of disease modifying agent within "delayed effect" 1 month of Visit 1 with: glucorticoids, cyclophosphamide, cyclosporine, cellcept
4. Therapies and/or medications:

   * History of previous use of Acthar for treatment of nephrotic syndrome
   * Prior sensitivity to Acthar or other porcine protein products
   * Planned treatment with live or live attenuated vaccines once enrolled in the study
5. Chronic systemic corticosteroid use, defined as any dose of systemic corticosteroid taken for more than 4 consecutive weeks within 1 month prior to Visit 1 (use of topical, inhaled, or intra-articular corticosteroids is allowed)
6. Planned treatment with live or live attenuated vaccines once enrolled in the study.
7. Contraindication to Acthar per Prescribing Information*
8. For the purpose of this study: history of peptic ulcer is defined as 6 months or less prior to Visit 1.
9. Renal target disease exclusions*
10. Out of control or severe hypertension
11. History of Systemic Lupus Erythematosus
12. Uncontrolled Type 1 or type 2 diabetes mellitus (prior diagnosis of gestational diabetes mellitus is not an exclusion)
13. History of Deep Vein Thrombosis (DVT) 6 months or less prior to Visit 1
14. Presence of renal vein thrombosis:

    * Known current diagnosis by ultrasound, magnetic resonance imaging (MRI) or computed tomography scan
    * Signs or symptoms consistent with occurrence of acute renal vein thrombosis (hematuria in combination with flank pain and >30% unexplained acute rise in serum creatinine) with renal vein thrombosis confirmed by ultrasound, MRI or computed tomography scan
15. Reproductive status:

    * Women who are pregnant
    * Women who are breastfeeding
    * Women of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period, as evaluated by the Investigator (women who are not of childbearing potential are those that have a history of hysterectomy, bilateral oophorectomy, or are postmenopausal with no history of menstrual flow for 12 months or more prior to Visit 1
16. Chronic active hepatitis C or B infection
17. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation or who are known to be positive for human immunodeficiency virus
18. Undergoing or have received therapy for solid tumor malignancy 5 years or less prior to Visit 1 (with the exception of treated and cured basal cell or treated and cured squamous cell carcinoma)
19. Undergoing or have received therapy for blood malignancy 5 years or less from Visit 1
20. Cardiovascular:

    * History of or active congestive heart failure (NYHA Functional Classification Class II through IV) on http://sscts.org/ClassificationHeartFailureNYHA.aspx

    OR
    * History of known dilated cardiomyopathy with left ventricular ejection fraction 30% or less

    OR
    * Occurrence of any of the following within 3 months of Visit 1:

      * Unstable angina
      * Myocardial infarction
      * Coronary artery bypass graft or percutaneous transluminal coronary angioplasty
      * Transient ischemic attack or cerebrovascular disease; or Unstable arrhythmia
21. Administration of any other investigational medication or participation in an interventional clinical research study within 30 days of Visit 1
22. Abuse of alcohol or other substance abuse within the 6 months prior to Visit 1 as determined by the Investigator
23. Subject is a participating Investigator, study coordinator, employee of an Investigator, or immediate family member of any of the aforementioned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
To assess final protein/creatinine ratio | 12 months

SECONDARY OUTCOMES:
Number of Inflammatory cells- change from baseline to 12 months to assess final kidney histology and disease activity index | 12 months
Percent of fibrosis (measured by trichrome staining) - change from baseline to 12 months to assess final kidney histology and disease activity index | 12 months
IgA level - change from baseline to 12 months to assess final kidney histology, disease activity index, and disease status. | 12 months
Amount of sclerosed glomeruli - change from baseline to 12 months to assess final kidney histology and disease activity index | 12 months
Serum Creatinine - change from baseline to 2 years to assess disease status. | 2 years
Albumin - change from baseline to 2 years to assess disease status. | 2 years
Aldosterone - change from baseline to 2 years to assess disease status. | 2 years
Cortisol - change from baseline to 2 years to assess disease status. | 2 years
Lipid Profile - change from baseline to 2 years to assess disease status. | 2 years
P/Cr - change from baseline to 2 years to assess disease status. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Sheikh-Hamad, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Harris Health System Smith Clinic or Ben Taub Hospital, Houston, Texas, United States